CLINICAL TRIAL: NCT06249893
Title: Doppler Ultrasound Pulse Detection in Out-of-Hospital Cardiac Arrest Patients: A Feasibility Study.
Brief Title: Feasibility of Doppler Ultrasound for Pulse Detection in Out-of-Hospital Cardiac Arrest Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Ludwig Boltzmann Institute Digital Health and Patient Safety (Other); Emergency Medical Service of Vienna (Unknown)
Responsible Party: Principal Investigator, Philipp Metelka, Dr., Resident, Medical University of Vienna
Other Study IDs: 1549/2023
Record Dates: First submitted 2024-01-02; First posted 2024-02-08 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Arrest, Out-Of-Hospital
Keywords: Cardiac Arrest; Out-Of-Hospital Cardiac Arrest; OHCA; Ultrasound; Point-Of-Care Ultrasound; POCUS; Pulse Check; POCUS Pulse Check; Doppler Ultrasound; Femoral Artery
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Included patients
  Interventions: Other: Point-of-care vascular ultrasound

INTERVENTIONS:
Other: Point-of-care vascular ultrasound — Point-of-care ultrasound will be used to image the femoral vessels and to perform a pulsed-wave doppler measurement of blood flow during chest compressions and during pauses for rhythm and manual pulse checks.

SUMMARY:
The goal of this prospective observational study is to investigate the feasibility of using doppler point-of-care ultrasound on the femoral artery with a portable device to assess the presence of a pulse in patients suffering from cardiac arrest in the out-of-hospital environment. The main question is how often researchers are successful in acquiring the necessary ultrasound signal in the out-of-hospital environment.

DETAILED DESCRIPTION:
In this prospective observational study, a dedicated research team will be dispatched to cardiac arrest patients treated in the prehospital environment by emergency medical services (EMS). The team will use a portable ultrasound device to identify the femoral artery and conduct a pulsed wave (PW) doppler measurement during chest compressions as well as during chest compression pauses for rhythm analysis and save the recorded images. These ultrasound pulse checks will be conducted in parallel with the normal treatment of the patient, including manual pulse checks, and will only be conducted if ultrasound is possible without interference in the resuscitation. All treatment decisions will rest with the treating EMS team.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest treated by EMS
* Minimum age of 18 years

Exclusion Criteria:

* Pregnancy or suspected pregnancy
* Disapproval of the treating EMS team
* Adults under legal guardianship
* Inability to perform femoral artery doppler ultrasound due to limited access to the patient and possible interference with the treating EMS team
* Inability to perform femoral artery doppler ultrasound due to injuries or anatomic abnormalities in the femoral region or necessary emergent medical interventions in the femoral region
* Decision to transfer the patient to the hospital with ongoing CPR for emergent procedures such as extracorporeal CPR before femoral artery doppler ultrasound could be attempted
* Inability to safely perform femoral artery doppler ultrasound due to environmental hazards

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population comprises non-pregnant adults suffering out-of-hospital cardiac arrest of any cause who are treated with CPR by emergency medical services.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Feasibility of femoral artery doppler ultrasound | During cardiac arrest, up to 45 minutes
  If an ultrasound image of the femoral artery of sufficient quality for Doppler ultrasound can be obtained, the primary outcome will be considered to be positive.

SECONDARY OUTCOMES:
Time until ultrasound signal acquisition | During cardiac arrest, up to 45 minutes
  The time until successful acquisition of the doppler ultrasound signal will be measured in 2-minute CPR-intervals and 30-second intervals (e.g. second CPR-interval, first 30 seconds).
Discordance between doppler ultrasound and manual pulse checks. | During cardiac arrest, up to 45 minutes
  The presence of a doppler ultrasound flow signal during rhythm analysis and the result of the manual pulse check that is performed in parallel by the treating EMS team will be evaluated and analyzed for discordance.
Correlation of the result of manual pulse checks with doppler peak systolic velocity | During cardiac arrest, up to 45 minutes
  The correlation of the result of manual pulse checks performed by the treating EMS team with the peak systolic velocity measured by doppler ultrasound will be analyzed.
Patient factors influencing probability of successful doppler ultrasound image acquisition | After cardiac arrest, through study completion (a maximum of 1 year)
  Patient factors sex, age, approximated bodyweight and suspected cause of cardiac arrest will be analyzed for correlation with successful doppler ultrasound image acquisition.
Inter-observer variability in determining the quality of the doppler ultrasound signal. | After cardiac arrest, through study completion (a maximum of 1 year)
  The sonographer on site will assess the quality of the acquired doppler ultrasound images, as well as two ultrasound experts who will be blinded to the performing sonographer. The difference between these assessments will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Metelka, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Emergency Medical Service of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided